CLINICAL TRIAL: NCT01298986
Title: Atrial Fibrillation Ablation The Hybrid Approach Versus Traditional Management
Acronym: AF
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: No subjects were ever enrolled.
Sponsor: Inova Health Care Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10.126 Hybrid AF
Record Dates: First submitted 2011-02-16; First posted 2011-02-18 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Ablation of Atrial Fibrillation
Keywords: atrial fibrillation ablation procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Pulmonary Vein Isolation (Active Comparator): Patients who have paroxysmal or persistent atrial fibrillation but whose left atrium is < /= 5.0
  Interventions: Procedure: Pulmonary vein isolation ablation procedure for atrial fibrillation
- Hybrid procedure for patients with a left atrium < /= 5.0 cm (Experimental): A combined procedure where the cardiac surgeon will place the ablation lesions on top of the heart and the electrophysiologist will place the lesions inside the heart. 3D mapping with be used to guide the procedure. The left atrial appendage will be surgically managed.
  Interventions: Procedure: Hybrid procedure for ablation of atrial fibrillation
- Cox Maze Procedure (Active Comparator): All lesions of the Cox Maze procedure will be completed as originally described by Dr. James Cox using crypthermia. Patients will be randomized if there left atrium is >5.0 cm but < 6.1 cm and are experiencing paroxysmal or persistent atrial fibrillation
  Interventions: Procedure: The Cox Maze Procedure for Ablation of Atrial Fibrillation
- Hybrid Procedure (Experimental): A collaborative approach between electrophysiologist and surgeons for patients with a left atrium <5.0 cm and < 6.1 cm where the surgeon will epicardially place the ablation lesions and the electrophysiologist will place the lesion lines endocardially. 3D mapping will be used and the left atrial appendage will be surgically managed.
  Interventions: Procedure: Hybrid Procedure for Left Atrium >5 cm but < 6.1 cm

INTERVENTIONS:
Procedure: Pulmonary vein isolation ablation procedure for atrial fibrillation — The catheters will be introduced to the right atrium using the femoral vein as an access. Following a trans-septal puncture, ablation catheters will be placed in the left atrium under appropriate imaging and anticoagulation conditions (Standard of care). Following the positioning of the ablation catheters in the left heart cavity ablation to achieve PVI and left atrial isthmus line are going to be performed. Following the appropriate protocol of mapping and AF induction the right sided isthmus is going to be ablated to achieve a flutter line ablation as well. Following the procedure and following the appropriate standard of care protocols, the catheter are going to be retrieved and the procedure will be concluded. The left atrial appendage will be managed surgically. All ablation lines will be placed according to their current standard of practice using radiofrequency ablation technology and based on CARTO mapping.
  Arms: Pulmonary Vein Isolation
Procedure: Hybrid procedure for ablation of atrial fibrillation — The endoscope will be passed though a small port in the right thoracic cavity to the beating heart. The pericardium will be opened, the coronary sinus transected. The ablation catheters will pass underneath the SVC and IVC establishing access to the transverse and oblique sinuses. A box lesion will be epicardially placed around the pulmonary veins using cryothermia. An additional lesion line will be placed from the box lesion to the left atrial appendage. The ablation catheter will be left in place to guide the EP physicians in placing the right and left atrial flutter lines using radiofrequency. Electromagnetic mapping using a CARTO system and measuring for conduction block of the pulmonary veins will be conducted by the EP's. A second small port will then placed in the left thoracic cavity and the pericardium on the left side will be opened and the left atrial appendage will be ablated with the use of a clip placed around the left atrial appendage and tightened.
  Arms: Hybrid procedure for patients with a left atrium < /= 5.0 cm
Procedure: The Cox Maze Procedure for Ablation of Atrial Fibrillation — A 7-cm incision is placed and the chest is entered through the 4th or 5th intercostal space. The femoral artery and femoral vein are cannulated. The pericardium is opened. Cardiopulmonary bypass is instituted. The right sided lesions are applied using 3 purse-strings that are placed over the right atrial free wall. The right and left atrial lesions are done using cryoablation using either nitrous oxide or Argon. Next the left atrium is entered through a standard atriotomy placed in the interatrial groove. The base of the left atrial appendage is cryoablated and connected to the left upper pulmonary vein. All four pulmonary veins are then encircled using multiple application of cryo. An endocardial cryolesion is then placed posteriorly down to the level of the mid-mitral valve annulus and an epicardial cryolesion is placed on the coronary sinus directly across the atrial wall from the endocardial lesion. The left atrial appendage is then surgically managed.
  Arms: Cox Maze Procedure
Procedure: Hybrid Procedure for Left Atrium >5 cm but < 6.1 cm — The endoscope will be passed though a small port in the right thoracic cavity to the beating heart. The pericardium will be opened, the coronary sinus transected. The ablation catheters will pass underneath the SVC and IVC establishing access to the transverse and oblique sinuses. A box lesion will be epicardially placed around the pulmonary veins using cryothermia. An additional lesion line will be placed from the box lesion to the left atrial appendage. The ablation catheter will be left in place to guide the EP physicians in placing the right and left atrial flutter lines using radiofrequency. Electromagnetic mapping using a CARTO system and measuring for conduction block of the pulmonary veins will be conducted by the EP's. A second small port will then placed in the left thoracic cavity and the pericardium on the left side will be opened and the left atrial appendage will be ablated with the use of a clip placed around the left atrial appendage and tightened.
  Arms: Hybrid Procedure

SUMMARY:
Rationale: To determine the most beneficial ablation methodology for individual patients with paroxysmal or persistent atrial fibrillation (defined by the Heart Rhythm Society) as surgeons and electrophysiologists work together on a convergent procedure (hybrid) to place the epicardial and endocardial ablation lines.

Objectives: Catheter and surgical ablation are being offered today to patients with drug refractory and symptomatic atrial fibrillation. This study is designed to assess the most efficient ablation approach in patients with paroxysmal and persistent atrial fibrillation. In patients with left atrium size of less than 5.0 cm, a Hybrid approach (pulmonary vein isolation performed surgically will be combined with right and left atrial flutter lines performed using a transcatheter approach) will be compared to percutaneous catheter ablation to isolate the pulmonary veins and apply the left and right atrial flutter lines with removal of LA appendage. In the group of patients with left atrial size 5.0-6.0 cm the Hybrid approach is going to be compared to the minimally invasive Cox-Maze III procedure.

Our hypotheses with regard to the rate of return to sinus rhythm off antiarrhythmic drugs at 6 months will demonstrate that the Hybrid approach is going to be a: superior to percutaneous catheter ablation in the less than 5 cm left atrial group and b: non-inferior when compared to the Cox-Maze III procedure in the 5-6 cm left atrial cm group.

We hypothesize that the safety of all procedures will show no differences and that there will be no differences in clinical complications between groups.

DETAILED DESCRIPTION:
Study Type: This is an experimental study in which patients who present with either paroxysmal or persistent atrial fibrillation will be randomized based on their left atrial size (≤ 5.0 or > 5.0 but < 6.1 cm) to receive a hybrid ablation approach vs percutaneous catheter where in both procedures ablation will include pulmonary vein isolation with a left and right atrial flutter line for patients with a left atrium ≤ 5.0 cm. and hybrid approach will be compared to the Cox Maze III procedure for patients with a left atrium > 5.0 < 6.1 cm .

Study Design: One hundred and fifty two patients (n=152) with persistent or paroxysmal atrial fibrillation who present for surgical or catheter ablation intervention are to be enrolled. The study will take place at the Inova Heart and Vascular Institute in Falls Church, VA in the specially designed hybrid surgical suite in the cardiovascular operating area. We expect enrollment to take (two years study duration). Patients will be included if they present for ablation with paroxysmal or persistent atrial fibrillation as defined by the Heart Rhythm Society and their left atrium is < 6.1 cm (volume). Patients will be excluded if they present with long standing persistent atrial fibrillation as defined by the Heart Rhythm Society, require other cardiac surgery, are unable to take anticoagulation or require prescribed anti arrhythmic medication for reason other than atrial fibrillation, have a left atrium measuring greater than 6.0 cm (volume),have had previous catheter ablation for atrial fibrillation (Do not exclude for prior AVNRT) or a pacemaker, are less than 18 years of age, are unable or unwilling to be followed according to set protocol to include implantation of a heart monitor 6 weeks prior to their ablation procedure.

Study Methodology: This is an experimental study in which patients who present with either paroxysmal or persistent atrial fibrillation will be randomized based on their left atrial size.

For patients with a left atrium size of less than 5.0 cm, a Hybrid approach (pulmonary vein isolation performed surgically will be combined with right and left atrial flutter lines performed using a transcatheter approach) will be compared to percutaneous catheter ablation to isolate the pulmonary veins and apply the left and right atrial flutter lines. In the group of patients with left atrial size of 5.0-6.0 cm the Hybrid approach is going to be compared to the minimally invasive Cox-Maze III procedure (Figure 1). Each patient regardless of procedure will have their left atrial appendage closed. All patients will receive an internal event monitor (Reveal XT) which will be placed 6 weeks before their procedure to establish atrial fibrillation burden. All patients will also be given a health related quality of life and a symptom frequency and severity tool to fill out prior to their ablation and at 3 and 6 months post ablation.

The primary outcome will be the rate of return to sinus rhythm as defined by the Heart Rhythm Society Guidelines (sinus rhythm maintained off anti arrhythmic medications and any monitored atrial arrhythmia greater than 30 seconds will be considered a recurrence) at 6 months and atrial fibrillation burden

The secondary outcomes will include:

Number and type of procedural complications Number of embolic strokes The number of major bleeding events as defined by the need to receive a transfusion for the amount of blood lost and or hemorrhagic stroke while receiving anticoagulation therapy.

Reported improvement in patients' self reported health related quality of life and their symptom frequency and severity at 3 and 6 months

Statistical Methodology: Since this is a proof of concept study without any prior literature to obtain margins, we used the current rate of return to sinus rhythm as our margins to determine sample size. This is fully explained in section 4.2. Based on these calculations, 152 patients will be randomized as described above. Descriptive statistics will be used to characterize the patient population. T-tests and ANOVAs will be used to look for differences between groups within the continuous data. Chi square, Fisher's Exact test and/or McNemar's Test will be used to look for differences among categorical variables. For all analyses, a two-sided p value <0.05 will be used to determine significance.

To analyze the primary objective, the percentage of patients in each group who return to normal sinus rhythm will be calculated. Chi square analysis, or logistic regression if covariates are required, will be used to test for differences in the odds of returning to normal sinus rhythm between the treatment groups in both arms of the study. Chi square and/or logistic regression will also be used to assess the secondary aim regarding complications between the treatment groups. For the left atrial size > 5.0 but < 6.1 cm arm of the study, testing for non-inferiority of complication rates will be conducted using the treatment effect and 95% confidence intervals. These will be compared against the 10% non-inferiority margins, to assess whether the treatment effect and 95% confidence interval fall entirely within the margins. Lastly, repeated measures analysis of variance (ANOVA) will be conducted to examine the secondary aim regarding change in health-related quality of life by treatment groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients will be included if they present for ablation with paroxysmal or persistent atrial fibrillation as defined by the Heart Rhythm Society and their left atrium is < 6.1 cm (volume)
2. Patients must be symptomatic with their AF as noted by their inability to perform their daily activities due to shortness of breath, fatigue, palpitations or other debilitating symptoms
3. Paroxysmal atrial fibrillation is defined as atrial fibrillation that resolves on its own within 7 days of onset
4. Persistent atrial fibrillation is defined as atrial fibrillation that does not resolve on its own and requires medical intervention to include medication therapy and/or electric cardioversion

Exclusion Criteria:

1. Patients will be excluded if they present with long standing persistent atrial fibrillation as defined by the Heart Rhythm Society
2. All patients with MV +2 mitral regurgitation will be excluded
3. Require other cardiac surgery procedures will be excluded
4. Are unable to take anticoagulation
5. Are unable to take any prescribed anti arrhythmic medication
6. Have a left atrium measuring greater than 6.0 cm (volume)
7. Have had previous catheter ablation for atrial fibrillation
8. Have had previous pace maker implantation
9. Are less than 18 years of age
10. Do not speak English and no translation can be provided
11. Are unable or unwilling to be followed according to set protocol to include obtaining an internally heart monitor 6 weeks prior to their ablation procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Return to sinus rhythm rate | 2-3 years
  The primary outcome will be the rate of return to sinus rhythm as defined by the Heart Rhythm Society Guidelines (sinus rhythm maintained off anti arrhythmic medications and any monitored atrial arrhythmia greater than 30 seconds will be considered a recurrence) at 6 months.

SECONDARY OUTCOMES:
Post procedure morbidities | up to 6 months post procedure
  The secondary outcomes will include:
  Total AF burden Number and type of procedural complications Number of embolic strokes The number of major bleeding as defined by the need to receive a transfusion for the amount of blood lost and or hemorrhagic stroke while receiving anticoagulation therapy.
  Reported improvement in patients' self reported health related quality of life and their symptom frequency and severity at 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Niv Ad, MD, Principal Investigator — Inova Fairfax Hospital